CLINICAL TRIAL: NCT06243133
Title: Pair Antiplatelet THerapy in Ischemic Stroke With Intracranial Artery Stenosis
Acronym: PATH-ICAS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Nengwei Yu, Head of neurology at Sichuan Provincial People's Hospital, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20223972
Record Dates: First submitted 2024-01-28; First posted 2024-02-06 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke; Intracranial Arteriosclerosis; Secondary Prevention; Antiplatelet Drug
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual antiplatelet therapy for 30 days (Experimental): Clopidogrel 300mg on the first day, then 75mg/ day for 30 consecutive days; Aspirin 100mg/ day for 90 days
  Interventions: Drug: clopidogrel for 30 days combined with aspirin for 90 days
- Dual antiplatelet therapy for 90 days (Active Comparator): Clopidogrel 300mg on the first day, then 75mg/day for 90 consecutive days; Aspirin 100mg/day for 90 days
  Interventions: Drug: clopidogrel for 90 days combined with aspirin for 90 days

INTERVENTIONS:
Drug: clopidogrel for 90 days combined with aspirin for 90 days — Clopidogrel 300mg on the first day, then 75mg/day for 90 consecutive days; Aspirin 100mg/day for 90 days
  Arms: Dual antiplatelet therapy for 90 days
Drug: clopidogrel for 30 days combined with aspirin for 90 days — Clopidogrel 300mg on the first day, then 75mg/ day for 30 consecutive days; Aspirin 100mg/ day for 90 days
  Arms: Dual antiplatelet therapy for 30 days

SUMMARY:
The goal of this clinical trial is to learn about efficacy and safety of dual antiplatelet therapy in ischemic stroke with intracranial artery stenosis. The main question it aims to answer are:

whether aspirin combined with clopidogrel for 3 month is better than 1 months for patients with non-cardiogenic cerebral infarction with intracranial artery stenosis.

Participants will get dual antiplatelet therapy (aspirin plus clopidogrel) for 1 month or 3 months within 7 days of the first stroke.

Researchers will compare experimental group (3 months dual antiplatelet therapy) with comparison group (1 month dual antiplatelet therapy), to see if experimental group would reduce stroke recurrence or mortality, and increase bleeding and other adverse prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 ~ 80 years old;
2. Patients diagnosed as non-cardiogenic cerebral infarction according to the WHO definition of stroke, with MRA/CTA/DSA confirmed intracranial artery stenosis ≥50% (intracranial carotid artery, M1 and proximal M2 segment of middle cerebral artery, A1 and A2 segment of anterior cerebral artery, P1 and P2 segment of posterior cerebral artery, intracranial vertebral artery and basilar artery);
3. First stroke onset within 7 days;
4. NIHSS score ≤5;
5. Patients or family members sign informed consent forms;

Exclusion Criteria:

1. Patients receiving thrombolysis or endovascular therapy;
2. Patients with recurrent stroke;
3. Patients has undergone major surgery or major trauma within the past 30 days;
4. History of gastrointestinal bleeding, active peptic ulcer, intracranial hemorrhage or other hemorrhagic diseases;
5. Contraindications or intolerances to the use of antiplatelet therapeutics;
6. Platelet count <100*109/L, hemoglobin<110g/L;
7. Patients with severe organ insufficiency or other serious disease (e.g., severe cardiopulmonary failure, advanced tumor, severe dementia);
8. Patients intolerant to MRI scan are replaced by CT or DSA;
9. poor compliance, unable to meet the requirements of the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
3-month major ischemic events and major bleeding events | 3-month
  Including any of the following: Cardiovascular and cerebrovascular mortality, Incidence of stroke (including ischemic and hemorrhagic), Incidence of myocardial infarction, bleeding events classified by BARC (Bleeding Academic Research Consortium) criteria

SECONDARY OUTCOMES:
disability | 3-month
  mRS(Modified Rankin Scale)>2
Cardiovascular or cerebrovascular mortality | 3-month
  mortality of Cardiovascular or cerebrovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Nengwei Yu, master, Study Chair — Sichuan Provincial People's Hospital; Jie Yang, doctor, Study Chair — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu S, Wu B, Liu M, Chen Z, Wang W, Anderson CS, Sandercock P, Wang Y, Huang Y, Cui L, Pu C, Jia J, Zhang T, Liu X, Zhang S, Xie P, Fan D, Ji X, Wong KL, Wang L; China Stroke Study Collaboration. Stroke in China: advances and challenges in epidemiology, prevention, and management. Lancet Neurol. 2019 Apr;18(4):394-405. doi: 10.1016/S1474-4422(18)30500-3. PMID 30878104
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Wang Y, Zhao X, Liu L, Soo YO, Pu Y, Pan Y, Wang Y, Zou X, Leung TW, Cai Y, Bai Q, Wu Y, Wang C, Pan X, Luo B, Wong KS; CICAS Study Group. Prevalence and outcomes of symptomatic intracranial large artery stenoses and occlusions in China: the Chinese Intracranial Atherosclerosis (CICAS) Study. Stroke. 2014 Mar;45(3):663-9. doi: 10.1161/STROKEAHA.113.003508. Epub 2014 Jan 30. PMID 24481975
- [Background] Wong KS, Chen C, Fu J, Chang HM, Suwanwela NC, Huang YN, Han Z, Tan KS, Ratanakorn D, Chollate P, Zhao Y, Koh A, Hao Q, Markus HS; CLAIR study investigators. Clopidogrel plus aspirin versus aspirin alone for reducing embolisation in patients with acute symptomatic cerebral or carotid artery stenosis (CLAIR study): a randomised, open-label, blinded-endpoint trial. Lancet Neurol. 2010 May;9(5):489-97. doi: 10.1016/S1474-4422(10)70060-0. Epub 2010 Mar 22. PMID 20335070
- [Background] Valgimigli M, Frigoli E, Heg D, Tijssen J, Juni P, Vranckx P, Ozaki Y, Morice MC, Chevalier B, Onuma Y, Windecker S, Tonino PAL, Roffi M, Lesiak M, Mahfoud F, Bartunek J, Hildick-Smith D, Colombo A, Stankovic G, Iniguez A, Schultz C, Kornowski R, Ong PJL, Alasnag M, Rodriguez AE, Moschovitis A, Laanmets P, Donahue M, Leonardi S, Smits PC; MASTER DAPT Investigators. Dual Antiplatelet Therapy after PCI in Patients at High Bleeding Risk. N Engl J Med. 2021 Oct 28;385(18):1643-1655. doi: 10.1056/NEJMoa2108749. Epub 2021 Aug 28. PMID 34449185
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Background] Johnston SC, Easton JD, Farrant M, Barsan W, Conwit RA, Elm JJ, Kim AS, Lindblad AS, Palesch YY; Clinical Research Collaboration, Neurological Emergencies Treatment Trials Network, and the POINT Investigators. Clopidogrel and Aspirin in Acute Ischemic Stroke and High-Risk TIA. N Engl J Med. 2018 Jul 19;379(3):215-225. doi: 10.1056/NEJMoa1800410. Epub 2018 May 16. PMID 29766750